CLINICAL TRIAL: NCT02018393
Title: Case-control Pilot Study of the Immune Modulating Effect of FEIBA on Patients
Brief Title: Case-control Pilot Study of the Immune Modulating Effect of FEIBA on Patients With Haemophilia A and Inhibitors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Victor Jimenez-Yuste, Medical Degree PhD, Hospital Universitario La Paz
Other Study IDs: PI-1405
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Severe Haemophilia A With Inhibitors
Keywords: FEIBA®

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Prophylaxis group: Prophylaxis with FEIBA is defined in this study as the regular infusion of FEIBA for the prevention of bleeding at a dose of ≥50 UF/kg on at least three non-consecutive days a week. Patients must have been on this modality for at least 6 months prior to the study visit
- On demand group: On-demand Treatment is defined as the administration of FEIBA only to control bleeding. Patients must have been on this modality for at least 6 months prior to the study visit.

SUMMARY:
This study aims to evaluate the immunomodulatory effect of FEIBA® in patients with severe haemophilia A and inhibitors.

DETAILED DESCRIPTION:
This is an observational, multicentric, case-control and one-single-visit study of patients with severe haemophilia A and inhibitors against FVIII in therapy with FEIBA®.

Two subject groups will be included: Group 1 (cases) will be composed of patients with severe haemophilia A and inhibitors in prophylaxis with FEIBA®; Group 2 (controls) will be composed of patients with severe haemophilia A and inhibitors on-demand treatment with FEIBA®.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has signed and dated the Informed Consent form for participation in this study.
2. Age ≥ 18 years old.
3. Patient with severe haemophilia A (FVIII <1%) and high-responding inhibitor (titre >5 UB) at some point in their life, currently on therapy with FEIBA® to control bleeding.
4. Group 1: Patients in prophylaxis with FEIBA®: The patient has been on prophylaxis regimen with FEIBA® for at least 6 months prior to the study visit. Group 2: Patients on-demand regimen with FEIBA®: The patient has been under on-demand treatment with FEIBA® for at 6 months prior to the study visit.

Exclusion Criteria:

1. The presence of any inflammatory condition at the time of the study visit or the previous 30 days that, according to the medical criterion, would affect the study objectives.
2. The patient is under immune tolerance treatment or has been at any time during the 30 days prior to the study visit.
3. The administration of any anti-inflammatory or immunosuppressive drug 15 days before the study visit.
4. Levels of CD4 <200/l regardless of the HIV status.
5. Altered hepatic or renal function defined by the presence of abnormal levels of alanine aminotransferase (ALAT) or serum creatinine, respectively.
6. Administration of any haemostatic treatment to control bleeding within the 5 days prior to the study visit.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe haemophilia A and inhibitors treated with FEIBA® (on demand or prophylaxis) for the control of bleedings.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of plasma levels of anti-FVIII antibodies (neutralising and non-neutralising) | At inclusion

SECONDARY OUTCOMES:
Measurement of the serum levels of inflammatory cytokines | At inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Victor Jimenez-Yuste, Medical doctor, PhD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- University Hospital La Paz, Madrid, Spain